CLINICAL TRIAL: NCT00583596
Title: Closure Of Patent Ductus Arteriosus With the AMPLATZER Duct Occluder the AMPLATZER® Duct Occluder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AGA-004; G980103
Expanded Access: NCT00583583 (No longer available)
Record Dates: First submitted 2007-12-20; First posted 2007-12-31 (Estimated); Results first posted 2014-07-18 (Estimated); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Patent Ductus Arteriosus (PDA)
Keywords: patent ductus arteriosus (PDA)
MeSH Terms: conditions — Ductus Arteriosus, Patent

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- implant to close PDA (Experimental)
  Interventions: Device: Device closure with AMPLATZER Duct Occluder; Other: Objective Performance Criteria

INTERVENTIONS:
Device: Device closure with AMPLATZER Duct Occluder — Device closure with AMPLATZER Duct Occluder
Other: Objective Performance Criteria — Compare results of device closure to objective performance criteria

SUMMARY:
AGA-004 - The objective of the study is to determine safety, effectiveness and clinical utility of the AMPLATZER Duct Occluder in patients with patent ductus arteriosus. AGA-007 - The objective of this study is to evaluate the long term safety and effectiveness issues that may not have have been adequately addressed during AGA-004.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a demonstrated patent ductus arteriosus
* Body weight > 5 Kilograms

Exclusion Criteria:

* Pulmonary vascular resistance above 8 Woods units or a Rp/Rs >0.4.
* Additional cardiac or non-cardiac abnormality that can reasonably be expected to significantly affect the patient's health adversely in the next two years, i.e.: cancer, Eisenmenger's syndrome, other serious congenital heart disease.
* Pelvic vein or inferior vena cava thrombosis
* Sepsis (local/generalized) or any type of infection that cannot be successfully treated prior to device placement.
* History of repeated pulmonary infection
* Demonstrated intracardiac thrombi on echocardiography • Inability to obtain informed consent

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 436 (Actual)
Dates: Start 1999-10; Primary Completion 2008-04 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (24):
- United States (24):
  - University of Alabama, Birmingham, Alabama
  - Children's Hospital, San Diego, California
  - Children's Hospital, Denver, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Florida, Gainesville, Florida
  - Arnold Palmer Hospital, Orlando, Florida
  - University of Chicago, Chicago, Illinois
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Louisana State University Medical Center, New Orleans, Louisiana
  - New England Medical Center, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Washington University Medical Center, St Louis, Missouri
  - Children's Hospital UN/CU), Omaha, Nebraska
  - Columbia University, New York, New York
  - Childrens Hospital, Rochester, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Texas, Dallas, Texas
  - Cook Children's Heart Center, Fort Worth, Texas
  - Children's Hospital of the King's Daughters, Norfolk, Virginia
  - University of Washington Medical Center, Seattle, Washington
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited in medical clinics. The first subject enrolled was September 10, 1999. The last follow-up occurred in the Post Market Surveillance Study on August 29, 2008.
Pre-assignment Details: Subjects meeting the inclusion/exclusion criteria of the protocol were included in the original clinical trial.
Groups:
- Long Term Follow-up for Subjects Implanted With the Device: Subjects enrolled in IDE study subject to Post Market Surveillance
Period: Overall Study
Arm/Group | Long Term Follow-up for Subjects Implanted With the Device
Started | 436 (Subjects in Phase 2 clinical trial who received the AMPLATZER Duct Occluder.)
Completed | 152
Not Completed | 284
Not completed — Lost to Follow-up | 110
Not completed — Excluded due to Hurricane Katrina | 30
Not completed — Death | 2
Not completed — Withdrawal by Subject | 6
Not completed — Lost to Follow-up | 94
Not completed — Data not complete | 1
Not completed — Not consented | 15
Not completed — Outside f-up window | 26

BASELINE CHARACTERISTICS:
Arm/Group | Long Term Follow-up for Subjects Implanted With the Device
Number analyzed (Participants) | 436
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.14 (11.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 298
  Male | 138
Region of Enrollment [Number; unit: participants]
  United States | 436

OUTCOME MEASURES:

1. Primary Outcome: Reporting of Late Adverse Events Relating to the Device.
Time Frame: Long term follow up for data captured at 5, 6 or 7 years post implant
Population: 152 subjects of the 436 subjects eligible for post market survelliance completed a 5, 6 or 7 year follow-up.
Measure: Number; unit: participant
Groups:
- Long Term Follow-up for Subjects Implanted With the Device: Subjects implanted with Amplatzer duct occluder that have final follow-up taking place 5 yrs., 6 yrs., or 7 yrs., post implant.
Arm/Group | Long Term Follow-up for Subjects Implanted With the Device
Number analyzed (Participants) | 152
participant | 9

2. Primary Outcome: Reporting of Late Efficacy Issues Regarding Patent Ductus Arteriosis (PDA) Closure
Description: The number of participants with a residual shunt (efficacy)
Time Frame: Long term follow up data captured at 5, 6 or 7 years post implant
Population: Of the 152 subjects that completed long term follow-up, 128 subjects underwent Transthoracic echocardiogram (TTE) at their final visit.
Measure: Number; unit: participants
Arm/Group | Long Term Follow-up for Subjects Implanted With the Device
Number analyzed (Participants) | 128
participants | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected during routine follow-up visits or if an event occurred between visits.
Arm/Group | Long Term Follow-up for Subjects Implanted With the Device
Serious Adverse Events (participants affected / at risk) | 1/436
Other Adverse Events (participants affected / at risk) | 8/436
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Long Term Follow-up for Subjects Implanted With the Device (N=436)
Obstruction of Pulmonary Artery with Gradient (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Long Term Follow-up for Subjects Implanted With the Device (N=436)
Mitral Valve regurgitation (Cardiac disorders) | 1 (1)
Left Pulmonary artery stenosis (Cardiac disorders) | 1 (1)
Aortic Stenosis with Chest Pain (Cardiac disorders) | 1 (1)
Death (General disorders) | 1 (1)
Atrial ectopic beats (Cardiac disorders) | 1 (1)
Echo finding (Cardiac disorders) | 1 (1)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Diabetic ketoacidosis (Endocrine disorders) | 1 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No